CLINICAL TRIAL: NCT05295290
Title: Low Interventional Cohort Study of Myocarditis/Pericarditis Associated With COMIRNATY in Persons Less Than 21 Years of Age
Brief Title: A Study to Learn About The COVID-19 (Study) Vaccine (Called COMIRNATY) in People That Are Less Than 21 Years Old.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Carelon Research (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C4591036
Record Dates: First submitted 2022-01-10; First posted 2022-03-25 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Myocarditis
Keywords: COMIRNATY; post-vaccine; COVID-19; MIS-C
MeSH Terms: conditions — Myocarditis; COVID-19

STUDY DESIGN:
Masking Description: This is a low-interventional cohort study to determine cardiac and non-cardiac long-term outcomes of persons less than 21 years of age with myocarditis/pericarditis after the administration of COMIRNATY, compared with similarly aged persons with myocarditis/pericarditis associated with COVID-19, including MIS-C, without exposure to COMIRNATY.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- myocarditis/pericarditis following COMIRNATY (Other): myocarditis/pericarditis following COMIRNATY within 28 days of dose
  Interventions: Diagnostic Test: Cardiac Imaging
- myocarditis/pericarditis following COVID-19 or MIS-C (Other): myocarditis/pericarditis following COVID-19 or MIS-C without exposure to COMIRNATY
  Interventions: Diagnostic Test: Cardiac Imaging

INTERVENTIONS:
Diagnostic Test: Cardiac Imaging — ECG, echocardiogram, ambulatory monitor, exercise stress test

SUMMARY:
The purpose of this clinical trial is to learn about the safety and effects of the study vaccine (called COMIRNATY) for the potential prevention of COVID-19. This study is seeking participants who:

1. Are age <21 years.
2. Have presentation to participating medical center with evaluation in Emergency Room and/or hospitalization.
3. Received either the 1st, 2nd, 3rd or booster dose(s) of COMIRNATY within 7 days of symptom onset.
4. Meet criteria of Centers for Disease Control and Prevention case definition of probable or confirmed myocarditis/pericarditis
5. Are capable of giving signed informed consent/assent (by parents/legal guardians of minors and/or patients), which includes compliance with the requirements and restrictions listed in the Informed Consent/Assent Document and in this protocol OR meets criteria for waiver of consent.

This study will examine the potential long-term effects associated with myocarditis/pericarditis following vaccination with COMIRNATY. The association of myocarditis/pericarditis in participants who received the study vaccine (COMIRNATY) compared with those associated with COVID-19 will also be examined. This will help us determine if COMIRNATY is safe and effective, and if there is a myocarditis/pericarditis association that should be noted. Participants will take part in this study for up to 5 years. During this time, they will receive complete cardiac imaging tests, and have follow up visits per guidance stated in the study protocol.

DETAILED DESCRIPTION:
This is a low-interventional cohort study to determine cardiac and non-cardiac long-term outcomes of persons <21 years of age with myocarditis/pericarditis after the administration of COMIRNATY, compared with similarly aged persons with myocarditis/pericarditis associated with COVID-19, including MIS-C.

To be classified as having COMIRNATY-associated myocarditis/pericarditis, a person must 1) meet the CDC case definition for probable or confirmed myocarditis/pericarditis, 2) have received any dose of COMIRNATY ≤ 7 days of symptom onset, and 3) have no other plausible alternative etiology at the time of enrollment.

To be classified as having myocarditis/pericarditis associated with COVID-19, a person must have 1) either acute severe COVID-19 infection or MIS-C, as defined by the CDC, 2) findings of probable or confirmed myocarditis in the CDC definition, 3) no other plausible alternative etiology. A description of the three cohorts is as follows:

Cohort 1: Prospectively ascertained cases of probable or confirmed myocarditis/pericarditis associated with COMIRNATY , i.e., participants enrolled under protocol during hospitalization or </= 2 weeks of hospital discharge.

Cohort 2: Retrospectively ascertained cases of probable or confirmed myocarditis/pericarditis associated with COMIRNATY , i.e., participants enrolled > 2 weeks after hospital discharge. Participants can be retrospectively ascertained and enrolled at any time from their COMIRNATY-associated myocarditis/pericarditis.

Cohort 3: Comparator cohort of COVID-19- related myocarditis/pericarditis , including MIS-C, both retrospectively and prospectively ascertained, and enrolled at any time from their COVID-19 or MIS-C associated myocarditis/pericarditis diagnosis.

Participants in all cohorts will be those who present to participating medical centers for care. This study is a collaboration between the National Heart, Lung, and Blood Institute (NHLBI)'s Pediatric Heart Network (PHN) and Pfizer.

Enrollment will include approximately 300 prospectively and retrospectively ascertained cases of children, adolescents, and young adults <21 years of age who receive care for myocarditis/pericarditis associated with COMIRNATY (Cohort 1 and 2); and approximately 100 persons <21 years of age with COVID -19-associated myocarditis/pericarditis, including MIS-C (Cohort 3).

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1/2:

  1. Age <21 years.
  2. Presentation to participating medical center with evaluation in Emergency Room and/or hospitalization.
  3. Received either the 1st, 2nd, 3rd or booster dose(s) of COMIRNATY within 28 days of symptom onset.
  4. Meets criteria of Centers for Disease Control and Prevention case definition of probable or confirmed myocarditis/pericarditis
  5. Capable of giving signed informed consent/assent (by parents/legal guardians of minors and/or patients), which includes compliance with the requirements and restrictions listed in the Informed Consent/Assent Document and in this protocol OR meets criteria for waiver of consent.
* Cohort 3:

  1. Age <21 years.
  2. Presentation to participating medical center with evaluation in Emergency Room and/or hospitalization.
  3. COVID-19-related disease

     1. Acute COVID-19 infection OR
     2. Multi-system Inflammatory Syndrome in Children Associated with COVID-19 (MIS-C) AND
  4. Probable or confirmed myocarditis/pericarditis* not temporally related to vaccination with COMINARTY

     1. Probable myocarditis/pericarditis as defined by ≥ 1 new finding of:

        * Elevated troponin above upper limit of normal
        * Abnormal ECG or rhythm monitoring finding consistent with myocarditis
        * Abnormal cardiac function or wall motion abnormalities on echocardiogram
        * cMRI findings consistent with myocarditis OR
     2. Confirmed myocarditis/pericarditis as defined by:

        * Histopathologic confirmation of myocarditis OR
        * Elevated troponin above upper limit of normal AND cMRI findings consistent with myocarditis
  5. Capable of giving signed informed consent/assent (by parents/legal guardians of minors and/or patients), which includes compliance with the requirements and restrictions listed in the Informed Consent/Assent Document and in this protocol OR meets criteria for waiver of consent.

Exclusion Criteria:

1. A plausible alternative etiology for myocarditis/pericarditis, as determined by the site based upon their routine clinical practice for evaluation of potential causes for myocarditis/pericarditis.
2. Pre-existing cardiac conditions that could impact the primary endpoint, including but not limited to, documented history of left ventricular dysfunction (e.g., cardiomyopathy or myocardial infarction), pacemaker, or congenital heart disease, with the exceptions of:

   1. Bicommissural aortic valve with < trivial stenosis and/or insufficiency
   2. Mitral valve prolapse with < trivial insufficiency
   3. Hemodynamically insignificant atrial septal or ventricular septal defects.
3. Previous administration with an investigational drug or vaccine within 30 days of enrollment (or as determined by the local requirement).

Ages: 0 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2030-11-21 (Estimated); Study Completion 2030-11-21 (Estimated)

PRIMARY OUTCOMES:
Composite findings of myocarditis | 6 months after illness onset
  This is a single composite primary outcome measure. This primary composite study endpoint is defined as the presence of 1 or more of the following 6 months after illness onset: left ventricular dysfunction (LVEF < 55% by echocardiogram), findings of myocarditis by original or revised Lake Louise criteria on cardiac MRI, or the presence of high-grade arrhythmia or conduction system disturbance on ECG or ambulatory monitoring.
Left ventricular ejection fraction (LVEF) < 55% by echocardiography | Up to 5 years following illness onset.
Myocarditis by original or revised Lake Louise criteria on cMRI | Up to 5 years following illness onset.
Arrhythmias on cardiac recording (ECG, ambulatory monitoring) | Up to 5 years following illness onset.
Complications, including non-cardiac morbidities by medical history | Up to 5 years following illness onset.
Functional Status by Behavior Assessment System for Children, Third Edition BASC-3 or PROMIS Short Forms | Up to 5 years following illness onset.
  Behavior Assessment System for Children, Third Edition (BASC-3), <8 yr (T score <30->70 with higher number meaning lower functioning) or PROMIS Short Forms ≥8 yr (scores from 3-15 with higher number meaning better functioning)
The Pediatric Quality of Life Inventory (PEDS QL) | Up to 5 years following illness onset.
  The 27 question, age-appropriate and parent-proxy questionnaires, will be used in 2 to <18-year-old participants to assess quality of life. Scores span 0-108 with higher number being better functioning.
The Quality of Life Scale (QOLS) | Up to 5 years following illness onset.
  The QOLS, a 16-item self-report form that assesses overall quality of life on a scale of 16-112 (higher scores indicate better quality of life) will be administered for participants ≥18 years old.
Conduction system disturbances on cardiac recording (ECG, ambulatory monitoring) | Up to 5 years following illness onset.

SECONDARY OUTCOMES:
Left ventricular ejection fraction (LVEF) by echocardiogram as a measure of myocardial performance. | During the hospitalization or within 2 weeks of hospital discharge, generally obtained less than 3 weeks from presentation.
Time to recovery of myocardial inflammation and injury by Lake Louise (the original or revised) criteria | During hospitalization or within 2 weeks of hospital discharge, commonly less than 3 weeks from presentation
Arrhythmias on cardiac recording (ECG, ambulatory monitoring) | During hospitalization or within 2 weeks of hospital discharge, commonly less than 3 weeks from presentation
Complications, including non-cardiac morbidities for myocarditis | During hospitalization or within 2 weeks of hospital discharge, commonly less than 3 weeks from presentation
Echocardiographic LVEF | Up to 5 years following illness onset.
Myocardial inflammation scarring (by cMRI) | Up to 5 years following illness onset.
Arrhythmias on cardiac recordings | Up to 5 years following illness onset.
Complications, including non-cardiac morbidities by medical history | Up to 5 years following illness onset.
Lower LVEF by composite results | Up to 5 years following illness onset.
  Identification of possible sociodemographic and medical risk factors for greater frequency and severity of acute and longer-term cardiac sequelae in participants, measured by ECG, original or revised Lake Louise criteria on cMRI, and presence of high-grade arrhythmia or conduction system disturbance on ECG or ambulatory monitoring.
For patients with isolated pericarditis, to determine time to recovery to normal. | At each study visit, up to 5 years, until the endpoint event is met
  Freedom from
  1. symptoms/signs of pericarditis;
  2. typical ECG findings of pericarditis;
  3. >small pericardial effusion;
  4. therapy with anti-inflammatory medications
Conduction system disturbances on cardiac recording (ECG, ambulatory monitoring) | During hospitalization or within 2 weeks of hospital discharge, commonly less than 3 weeks from presentation
Conduction system disturbances on cardiac recordings | Up to 5 years following illness onset.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (34):
- United States (33):
  - Children's of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Lucile Packard Children's Hospital Stanford, Palo Alto, California
  - Childrens Hospital of Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Nemours Children's Hospital, Delaware, Wilmington, Delaware
  - Childrens National Hospital, Washington D.C., District of Columbia
  - Memorial Healthcare System, Hollywood, Florida
  - Children's Healthcare of Atlanta - Arthur M. Blank Hospital, Atlanta, Georgia
  - Lurie Children's Hospital, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Riley Hospital for Children at IU Health, Indianapolis, Indiana
  - Children's Hospital, New Orleans, Louisiana
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan Health Center, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Children'S Hospitals & Clinics of Minn, Minneapolis, Minnesota
  - Childrens Mercy Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Northwell Health-Cohen Children's Medical Center, New Hyde Park, New York
  - Columbia University Medical Center, New York, New York
  - Duke University Hospital, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina: Shawn Jenkins Women's and Children's Hospital, Charleston, South Carolina
  - MUSC Summey Medical Pavilion, North Charleston, South Carolina
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4591036